CLINICAL TRIAL: NCT00529139
Title: The Hannover-Dialysis-Outcome (HAN-D-OUT)-Study: Comparison of Standard Versus Intensified Extended Dialysis in Treatment of Patients With Acute Kidney Injury in the Intensive-Care Unit
Brief Title: Hannover Dialysis Outcome Study
Acronym: HAND-OUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Fresenius AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHH - SLED - 01
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Acute Kidney Failure
Keywords: Extended dialysis; Acute kidney injury; Intensive care unit; Renal replacement therapy; Survival; Dialysis
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Device: Standard extended dialysis
- B (Active Comparator)
  Interventions: Device: Intensified extended dialysis

INTERVENTIONS:
Device: Standard extended dialysis — Standard extended dialysis dosed to maintain plasma urea levels between 120-150 mg/dL (20 -25 mmol/L)
  Arms: A
Device: Intensified extended dialysis — Intensified extended dialysis dosed to maintain near-normal plasma urea levels, i.e. <90 mg/dL (<15 mmol/L)
  Arms: B

SUMMARY:
Mortality rates of patients with acute kidney injury in the intensive care unit have changed little over the past few decades despite significant advances in supportive care. Few interventions have been shown to result in an improvement of in-hospital mortality of these patients, with dose of renal replacement therapy (RRT) being one of the most important. Patients undergoing continuous veno-venous hemofiltration had better outcomes with ultrafiltration rates of 35 mL/kg/h or 45 mL/kg/h than those treated at a rate of 20 mL/kg/h. In a different trial, intermittent hemodialysis on a daily basis resulted in better control of uremia, fewer hypotensive episodes during dialysis, and more rapid resolution of acute renal failure than thrice weekly hemodialysis. In the present study we examine survival and renal recovery in critically ill patients with acute kidney injury that are treated with a currently recommended (standard) dose of RRT, and patients that receive intensified RRT.

ELIGIBILITY:
Inclusion Criteria:

* non post-renal AKI with RRT dependency indicated by oliguria/anuria <30mL/h >6 hours prior to inclusion
* loss of kidney function of >30% within 48 hours prior to inclusion
* hyperkalemia >6.5 mmol/L
* severe acidosis with pH<7.15

Exclusion Criteria:

* pre-existing chronic kidney disease (CKD) as defined by an estimated glomerular filtration rate <50mL/min or a plasma creatinine concentration >1.7 mg/dL (>150 µmol/L) more than 10 days prior to initiation of the first RRT
* presence of AV-fistula or dialysis catheter
* participation in another study
* consent denial or withdrawal
* need for extra corporal membrane oxygenation therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2003-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Survival | Day 14 after initiation of renal replacement therapy

SECONDARY OUTCOMES:
Survival and renal recovery | Day 28 after initiation of renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Fliser, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Ghosh CC, Thamm K, Berghelli AV, Schrimpf C, Maski MR, Abid T, Milam KE, Rajakumar A, Santel A, Kielstein JT, Ahmed A, Thickett D, Wang K, Chase M, Donnino MW, Aird WC, Haller H, David S, Parikh SM. Drug Repurposing Screen Identifies Foxo1-Dependent Angiopoietin-2 Regulation in Sepsis. Crit Care Med. 2015 Jul;43(7):e230-40. doi: 10.1097/CCM.0000000000000993. PMID 25855898